CLINICAL TRIAL: NCT06984107
Title: Intra-operative Application of Polynucleotides-Hyaluronic Acid Hydrogel (Regenfast®) for the Surgical Treatment of Medication-related Osteonecrosis of the Jaws (MRONJ): a Pilot Study
Brief Title: MRONJ and Polynucleotides-Hyaluronic Acid Hydrogel (Regenfast®)
Acronym: REG-MRONJ-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7475
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Medication Related Osteonecrosis of the Jaw

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical resection plus polynucleotides and hyaluronic acid (PN+HA) (Experimental): Surgical management will be performed by reflecting a full-thick flap to expose the entire affected area, followed by removal of necrotic bone until a vital, unaffected bony margin will be obtained. After bone resection, the PN+HA (Regenfast®) will be applied on the residual bone surface. Wound management will be done via primary closure.
  Interventions: Device: MRONJ resection plus PN+HA

INTERVENTIONS:
Device: MRONJ resection plus PN+HA — Surgical management will be performed by reflecting a full-thick flap to expose the entire affected area, followed by removal of necrotic bone until a vital, unaffected bony margin will be obtained. After bone resection, the PN+HA (Regenfast®) will be applied on the residual bone surface. Wound management will be done via primary closure.

SUMMARY:
Several circumstances or conditions, such as wound extension or disease, can affect the hard and soft tissue healing after surgical treatment of MRONJ. Supportive therapies are therefore needed to help tissues wound healing. The primary objective of this pilot clinical case series is to evaluate the post-operative wound healing in a group of patients undergoing surgical therapy for MRONJ with intraoperative application of a gel based on polynucleotides and hyaluronic acid (PN+HA) (Regenfast®)

ELIGIBILITY:
Inclusion criteria:

* Patients older than 18 years
* Provided informed consent
* MRONJ stage 1 and stage 2 diagnosis, in accordance to SICMF-SIPMO classification
* Need to undergo surgical treatment of MRONJ

Exclusion criteria:

* Patients with history of head and neck radiotherapy
* Neurological and psychiatric conditions
* Pregnancy
* MRONJ stage 3 diagnosis
* Patients who will receive a re-treatment for MRONJ
* Patients with general contraindication for oral surgery
* Patients unable to attend the out-patients visits scheduled by the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical wound healing (modified Landry Healing Index) | 7 days after surgical treatment
  The clinical wound healing of the site will be assessed throughout the modified Landry Healing Index
Clinical wound healing (modified Landry Healing Index) | 14 days after surgical treatment
  The clinical wound healing of the site will be assessed throughout the modified Landry Healing Index
Clinical wound healing (modified Landry Healing Index) | 21 days after surgical treatment
  The clinical wound healing of the site will be assessed throughout the modified Landry Healing Index
Clinical wound healing (modified Landry Healing Index) | 3 months after surgical treatment
  The clinical wound healing of the site will be assessed throughout the modified Landry Healing Index
Clinical wound healing (modified Landry Healing Index) | 6 months after surgical treatment
  The clinical wound healing of the site will be assessed throughout the modified Landry Healing Index
Clinical wound healing (modified Landry Healing Index) | 12 months after surgical treatment
  The clinical wound healing of the site will be assessed throughout the modified Landry Healing Index

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Lajolo, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS